CLINICAL TRIAL: NCT04366310
Title: Capillary Refill Index Measurement with a Temperature Control Procedure
Brief Title: Capillary Refill Index with Rewarming
Acronym: CRI
Status: Terminated | Type: Observational
Why Stopped: Insufficient enrollment to achieve outcomes
Sponsor: Nihon Kohden (Industry)
Responsible Party: Sponsor
Other Study IDs: A960-055244; 20-0310 (Other: North Shore-Long Island Jewish Health System)
Record Dates: First submitted 2020-04-20; First posted 2020-04-28 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Peripheral Perfusion
Keywords: capillary refill time; peripheral perfusion
MeSH Terms: interventions — Rewarming

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- capillary refill index (CRI): a waveform analysis method using a pulse oximeter to assess peripheral perfusion
  Interventions: Device: capillary refill index; Procedure: rewarming

INTERVENTIONS:
Device: capillary refill index — a waveform analysis method using a pulse oximeter to assess peripheral perfusion
  Other Names: CRI
Procedure: rewarming — warming fingertip skin temperature using an instant hot pack

SUMMARY:
A new technology, capillary refill index (CRI) can be useful for assessing peripheral perfusion status quantitatively, but this value can be influenced by fingertip temperature. The aim of this study is to evaluate the predictive accuracy of CRI after a temperature control (warming) procedure in predicting 30-day mortality among ICU/CCU patients. The investigators hypothesized that lowered fingertip temperature can lead prolonged CRI values which are considered as false positives in detection of high-risk patients for mortality, because it causes poor peripheral perfusion which does not reflect hemodynamic instability. The investigators will use the warming procedure to remove or reduce the effect of the fingertip temperature on the CRI measurement and will analyze whether it contributes to reduction of false positives in detection of high-risk patients for mortality.

DETAILED DESCRIPTION:
Capillary refill time (CRT) test is a simple and noninvasive method typically used to assess peripheral blood perfusion at the bedside. CRT is defined as the time required for a distal capillary bed (e.g., fingertip) to regain its color after having received enough compression to cause blanching [1]. Because a prolonged CRT suggests a decrease in peripheral perfusion and poor peripheral perfusion is strongly associated with patients' mortality, several studies reported the clinical usefulness of CRT for predicting patients' mortality in the critical care setting [2,3]. However, because the conventional CRT test depends on clinicians' subjective visual assessment, the inter-rater agreement of it has been questioned, and substantial clinical experience is needed to acquire the reliable skill to measure CRT [4, 5, 6, 7]. Therefore, there is great demand for the creation of objective methods to easily assess peripheral blood perfusion.

Previously, the investigators developed a new mechanical device by using pulse oximetry waveforms, which can enable us to measure CRT easily and objectively. The measurement obtained with this device is called Capillary Refill Index (CRI) to differentiate it from traditional visual assessment of CRT [8]. The method calculates the time it takes for blood to return to the fingertip after release from compression by algorithmically analyzing the light intensity waveform of a normal pulse oximeter sensor attached to a patient's fingertip. The investigators' previous study showed that CRI can be an alternative to traditional CRT for assessing peripheral blood perfusion [8, 9, 10].

In the investigators previous study with healthy volunteer subjects [11], the investigators found that lowered fingertip temperature is a critical component that affects measurement values of CRI, which is the same phenomena with the traditional CRT. Since lowered skin temperature causes poor peripheral perfusion, the patients with lower fingertip temperature can show prolonged CRI without reflecting hemodynamic instability, which means lower skin temperature can increase false positives when using CRI to detect patients at high risk for mortality. The investigators hypothesize that the predictive accuracy of CRI for detecting patients at increased risk for mortality may be improved if the patients' skin temperature is warmed up before the measurement.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Admitted to any ICU of North Shore University Hospital (NSUH) within 24 hours

Exclusion Criteria:

* Pregnant
* Prisoners
* Finger, hand or forearm anatomical anomaly or disease that may interfere with attaching a pulse oximeter sensor
* Patients who are not deemed clinically stable by the clinical team
* Wearing nail polish, nail gel, or nail decorations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult intensive care unit (ICU) patients (both males and females without regards to ethnic and racial backgrounds)
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
AUC of ROC curve for 30 days mortality | 31 days
  Receiver operator characteristic (ROC) curve analysis of CRI after the temperature control procedure for 30 days mortality of ICU patients will be performed and area under the curve (AUC) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Timmy Li, PhD, Principal Investigator — Administrative Director Clinical Research Emergency Medicine, Northwell Health
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schriger DL, Baraff L. Defining normal capillary refill: variation with age, sex, and temperature. Ann Emerg Med. 1988 Sep;17(9):932-5. doi: 10.1016/s0196-0644(88)80675-9. PMID 3415066
- [Background] Lima A, Jansen TC, van Bommel J, Ince C, Bakker J. The prognostic value of the subjective assessment of peripheral perfusion in critically ill patients. Crit Care Med. 2009 Mar;37(3):934-8. doi: 10.1097/CCM.0b013e31819869db. PMID 19237899
- [Background] Ait-Oufella H, Bige N, Boelle PY, Pichereau C, Alves M, Bertinchamp R, Baudel JL, Galbois A, Maury E, Guidet B. Capillary refill time exploration during septic shock. Intensive Care Med. 2014 Jul;40(7):958-64. doi: 10.1007/s00134-014-3326-4. Epub 2014 May 9. PMID 24811942
- [Background] van Genderen ME, Paauwe J, de Jonge J, van der Valk RJ, Lima A, Bakker J, van Bommel J. Clinical assessment of peripheral perfusion to predict postoperative complications after major abdominal surgery early: a prospective observational study in adults. Crit Care. 2014 Jun 3;18(3):R114. doi: 10.1186/cc13905. PMID 24894892
- [Background] Alsma J, van Saase JLCM, Nanayakkara PWB, Schouten WEMI, Baten A, Bauer MP, Holleman F, Ligtenberg JJM, Stassen PM, Kaasjager KHAH, Haak HR, Bosch FH, Schuit SCE; FAMOUS Study Group*. The Power of Flash Mob Research: Conducting a Nationwide Observational Clinical Study on Capillary Refill Time in a Single Day. Chest. 2017 May;151(5):1106-1113. doi: 10.1016/j.chest.2016.11.035. Epub 2016 Dec 7. PMID 27940191
- [Background] Pickard A, Karlen W, Ansermino JM. Capillary refill time: is it still a useful clinical sign? Anesth Analg. 2011 Jul;113(1):120-3. doi: 10.1213/ANE.0b013e31821569f9. Epub 2011 Apr 25. PMID 21519051
- [Background] Shinozaki K, Jacobson LS, Saeki K, Kobayashi N, Weisner S, Falotico JM, Li T, Kim J, Lampe JW, Becker LB. Does training level affect the accuracy of visual assessment of capillary refill time? Crit Care. 2019 May 6;23(1):157. doi: 10.1186/s13054-019-2444-3. No abstract available. PMID 31060576
- [Background] Shinozaki K, Saeki K, Jacobson LS, Falotico JM, Li T, Hirahara H, Horie K, Kobayashi N, Weisner S, Lampe JW, Becker LB. Evaluation of accuracy of capillary refill index with pneumatic fingertip compression. J Clin Monit Comput. 2021 Feb;35(1):135-145. doi: 10.1007/s10877-019-00454-1. Epub 2020 Jan 8. PMID 31916222
- [Background] Shinozaki K, Capilupi MJ, Saeki K, Hirahara H, Horie K, Kobayashi N, Weisner S, Kim J, Lampe JW, Becker LB. Blood refill time: Clinical bedside monitoring of peripheral blood perfusion using pulse oximetry sensor and mechanical compression. Am J Emerg Med. 2018 Dec;36(12):2310-2312. doi: 10.1016/j.ajem.2018.04.006. Epub 2018 Apr 5. No abstract available. PMID 29678295
- [Background] Shinozaki K, Jacobson LS, Saeki K, Hirahara H, Kobayashi N, Weisner S, Falotico JM, Li T, Kim J, Becker LB. Comparison of point-of-care peripheral perfusion assessment using pulse oximetry sensor with manual capillary refill time: clinical pilot study in the emergency department. J Intensive Care. 2019 Nov 27;7:52. doi: 10.1186/s40560-019-0406-0. eCollection 2019. PMID 31798887
- [Background] Shinozaki K, Capilupi MJ, Saeki K, Hirahara H, Horie K, Kobayashi N, Weisner S, Kim J, Lampe JW, Becker LB. Low temperature increases capillary blood refill time following mechanical fingertip compression of healthy volunteers: prospective cohort study. J Clin Monit Comput. 2019 Apr;33(2):259-267. doi: 10.1007/s10877-018-0159-7. Epub 2018 May 30. PMID 29846867